CLINICAL TRIAL: NCT06256276
Title: Nutritional Therapy for Autonomic Dysfunction in Elderly Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 202617
Record Dates: First submitted 2024-02-02; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Carnitine; Psyllium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whey protein powder and L-carnitine capsules (Experimental): Subjects will daily consume whey protein powder to supplement normal daily protein intake up to 1.2g protein/kg body weight per day (1 or 2 scoops powder), as well as 2 capsules (1 gram) L-carnitine for 16 weeks.
  Interventions: Dietary Supplement: Whey protein powder and L-carnitine
- Maltodextrin placebo powder and Psyllium Husk capsules (Placebo Comparator): Subjects will daily consume maltodextrin powder as if to supplement normal daily protein intake up to 1.2g protein/kg body weight per day (1 or 2 scoops powder), as well as 2 capsules (1 gram) psyllium husk for 16 weeks.
  Interventions: Dietary Supplement: Maltodextrin placebo powder and Psyllium Husk capsules

INTERVENTIONS:
Dietary Supplement: Whey protein powder and L-carnitine — Dietary supplement intervention for 16 weeks
  Other Names: Dymatize Elite Whey, Europa Sports Products
  Arms: Whey protein powder and L-carnitine capsules
Dietary Supplement: Maltodextrin placebo powder and Psyllium Husk capsules — Maltodextrin placebo powder and Psyllium Husk capsules
  Arms: Maltodextrin placebo powder and Psyllium Husk capsules

SUMMARY:
Recent studies suggest that patients with heart failure (HF) may have a reduced ability to control the tone of their blood vessels, heart rate or blood pressure in response to stress. This study will test whether 16 weeks of protein supplements can improve control of blood pressure and heart rate in HF patients.

DETAILED DESCRIPTION:
Heart Failure is defined as "a complex clinical syndrome that can result from any structural or functional cardiac disorder that impairs the ability of the ventricle to fill or eject blood." The New York Heart Association classifies heart failure four functional classes: NYHA 1-4, with Class 1 as minimal and Class 4 as the most advanced stage.

As a clinical syndrome, HF can be associated with significant limitations in functional capacity which can be very debilitating in the elderly population. It is a major cause of morbidity and mortality and is the leading cause of hospitalization among older individuals in the United States (1-15), particularly among those aged ≥65 years (16, 18). Nearly 1 million hospitalizations for HF occur each year with rates of hospitalization continuing to rise. Prevalence of heart failure was estimated to be more than 5.8 million in the United States and HF was singled out as an emerging epidemic (17).

Heart failure is associated with autonomic and endothelial dysfunction. Recent studies suggest that patients with HF maybe more prone to having impaired vasomotor and autonomic response to stress (19-29). A reduced ability to increase blood flow or heart rate appropriately in response to demand could limit the functional capacity of these subjects and would contribute to orthostasis (drop in blood pressure on standing). Another factor contributing to orthostasis in these individuals is poor muscle tone in the lower extremities reducing venous flow.

Endothelial dysfunction in HF on the other hand is attributed to decreased production of NO and increased oxidative stress due to neurohumoral activation, release of inflammatory messengers from the myocardium, altered local shear force and resultant atherogenesis (30, 31). The endothelial dysfunction itself causes an increase in the production of cytokines, uncoupling of eNOS and further increases the oxidative stress (32-35). The endothelium helps in regulating the vascular tone by balancing the production of vasodilators and vasoconstrictors in response to various stimuli (36) and its dysfunction would also impair baroreceptor function which in turn would affect cardiac autonomic activity and blood flow.

In our research we hope to improve both autonomic and endothelial function by supplementing protein and carnitine in diet. Studies have shown that when protein is metabolized to the amino acids L-arginine and citrulline, there is increased synthesis of NO (37). L-arginine, a semi-essential basic amino acid, is a precursor in the formation of nitric oxide by the enzyme nitric oxide synthase and directly increases the formation of NO (38). The administration of arginine and/or citrulline in patients in HF has been reported to improve endothelial function. Systolic and diastolic arterial pressures as well as pulmonary arterial systolic pressure have been shown to decrease significantly after administration of arginine or citrulline administration, which in turn improves right ventricular diastolic diameter (37, 39). One clinical study reported improvement in pulmonary artery pressure and right ventricular ejection fraction after two months of oral supplementation with L-arginine or citrulline in patients with HF and right ventricular dysfunction (39). It is hoped that protein supplementation will improve autonomic function by having a positive impact on physiological and biochemical parameters, including nitric oxide synthesis which is expect will improve baroreceptor blood flow, autonomic BP and HR in response to tilt.

Carnitine supplementation of 1g/d for 12 wk in hemodialysis patients significantly reduced systemic inflammation, as reflected by decreases in CRP, IL-1β, and IL-6 (40). In obesity, the mitochondrial abnormalities of reduced fatty acid oxidation, incomplete β-oxidation, and impaired substrate switching from fatty acid to pyruvate were reversed after 8wks of oral supplementation with the same dosage of carnitine (41). It is anticipated the same beneficial effects of carnitine in individuals with HF.

The purpose of this study is to evaluate the effects of 16 weeks of protein supplementation on measures of autonomic regulation of blood pressure and heart rate, as well as physical strength and function in elderly subjects with mild to moderate heart failure (NYHA 1, 2, or 3). Each participant will be randomized to one of two groups (whey protein + L-carnitine or placebos). Study endpoints will be measured at baseline and after 4 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate heart failure (NYHA I, II, or III symptomology) as confirmed by study physician

Exclusion Criteria:

* Moderately-severe dementia (MoCA score)
* Active inflammatory bowel disease
* Active cancer or chemotherapy in the past year
* Self-reported allergy to whey protein
* Documented insulin-dependent diabetes mellitus, or uncontrolled diabetes with hemoglobin A1C >8.5% (collected from medical record)
* >50mg doses of metoprolol or atenolol daily or more than 12.5mg twice daily of carvedilol
* History of renal failure stage IV or V
* History of severe orthostasis (>20mm Hg drop in systolic pressure)
* History of high grade second degree heart block
* History of arrhythmias (atrial or ventricular, tachy or brady)
* Other criteria as determined by the study physician

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular assessment of blood pressure | Change from baseline to 16 weeks
  Measuring orthostatic blood pressure
Cardiovascular assessment | Change from baseline to 16 weeks
  Measuring heart rate before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gohar Azhar, M.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No